CLINICAL TRIAL: NCT06867406
Title: A Phase I, Single-Center, Open-Label Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of KPC000154 Tablets in Healthy Adult Volunteers
Brief Title: A Trial to Evaluate KPC000154 Tablets in Healthy Subjects
Acronym: KPC000154
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kunming Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPC000154-C101; kyjtcrc (Registry Identifier: Duo Gao)
Record Dates: First submitted 2025-02-27; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-12

CONDITIONS: Healthy Subjects、Lipid Metabolism

STUDY DESIGN:
Intervention Model Description: 1.To determine the pharmacokinetic profile and its variability of KPC000154 tablets after single oral administration in healthy subjects. 2.To determine the pharmacokinetic profile and its variability of KPC000154 tablets after multiple oral administrations in healthy subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Placebo (SAD) (Placebo Comparator): A placebo used in a single-dose study where participants receive either the experimental drug or the placebo.
  Interventions: Drug: Placebo-controlled（SAD）
- Placebo (MAD） (Placebo Comparator): A placebo used in a single-dose study where participants receive either the experimental drug or the placebo.
  Interventions: Drug: Placebo-controlled（MAD）
- KPC000154 10mg Tablet Intervention (Experimental): KPC000154, a thyroid hormone receptor beta (THR-β) agonist, is an investigational drug aimed at evaluating the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single 10 mg oral dose of KPC000154 tablets in healthy subjects.
  Interventions: Drug: KPC000154 10mg Tablet Intervention
- KPC000154 30mg Tablet Intervention (Experimental): KPC000154, a thyroid hormone receptor beta (THR-β) agonist, is an investigational drug aimed at evaluating the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single 10 mg oral dose of KPC000154 tablets in healthy subjects.
  Interventions: Drug: KPC000154 30mg Tablet Intervention
- KPC000154 60mg Tablet Intervention (Experimental): KPC000154, a thyroid hormone receptor beta (THR-β) agonist, is an investigational drug aimed at evaluating the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single 10 mg oral dose of KPC000154 tablets in healthy subjects.
  Interventions: Drug: KPC000154 60mg Tablet Intervention
- KPC000154 120mg Tablet Intervention (Experimental): KPC000154, a thyroid hormone receptor beta (THR-β) agonist, is an investigational drug aimed at evaluating the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single 10 mg oral dose of KPC000154 tablets in healthy subjects.
  Interventions: Drug: KPC000154 120mg Tablet Intervention
- KPC000154 200mg Tablet Intervention (Experimental): KPC000154, a thyroid hormone receptor beta (THR-β) agonist, is an investigational drug aimed at evaluating the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single 10 mg oral dose of KPC000154 tablets in healthy subjects.
  Interventions: Drug: KPC000154 200mg Tablet Intervention
- KPC000154 300mg Tablet Intervention (Experimental): KPC000154, a thyroid hormone receptor beta (THR-β) agonist, is an investigational drug aimed at evaluating the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single 10 mg oral dose of KPC000154 tablets in healthy subjects.
  Interventions: Drug: KPC000154 300mg Tablet Intervention
- KPC000154 400mg Tablet Intervention (Experimental): KPC000154, a thyroid hormone receptor beta (THR-β) agonist, is an investigational drug aimed at evaluating the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single 10 mg oral dose of KPC000154 tablets in healthy subjects.
  Interventions: Drug: KPC000154 400mg Tablet Intervention
- KPC000154 40mg multiple-dose Tablet Intervention（To Be Determined） (Experimental): Multiple doses of KPC000154 will be administered to healthy subjects to assess safety, tolerability, pharmacokinetics, and pharmacodynamics.
  Interventions: Drug: KPC000154 40mg multiple-dose Tablet Intervention（To Be Determined）
- KPC000154 80mg multiple-dose Tablet Intervention（To Be Determined） (Experimental): Multiple doses of KPC000154 will be administered to healthy subjects to assess safety, tolerability, pharmacokinetics, and pharmacodynamics.
  Interventions: Drug: KPC000154 80mg multiple-dose Tablet Intervention（To Be Determined）
- KPC000154 120mg multiple-dose Tablet Intervention（To Be Determined） (Experimental)
  Interventions: Drug: KPC000154 120mg multiple-dose Tablet Intervention（To Be Determined）

INTERVENTIONS:
Drug: KPC000154 10mg Tablet Intervention — KPC000154 10mg Tablet administered orally in the morning once daily for 1 day
  Arms: KPC000154 10mg Tablet Intervention
Drug: KPC000154 30mg Tablet Intervention — KPC000154 30mg Tablet administered orally in the morning once daily for 1 day
  Arms: KPC000154 30mg Tablet Intervention
Drug: KPC000154 60mg Tablet Intervention — KPC000154 60mg Tablet administered orally in the morning once daily for 1 day
  Arms: KPC000154 60mg Tablet Intervention
Drug: KPC000154 120mg Tablet Intervention — KPC000154 120mg Tablet administered orally in the morning once daily for 1 day
  Arms: KPC000154 120mg Tablet Intervention
Drug: KPC000154 200mg Tablet Intervention — KPC000154 200mg Tablet administered orally in the morning once daily for 1 day
  Arms: KPC000154 200mg Tablet Intervention
Drug: KPC000154 300mg Tablet Intervention — KPC000154 300mg Tablet administered orally in the morning once daily for 1 day
  Arms: KPC000154 300mg Tablet Intervention
Drug: KPC000154 400mg Tablet Intervention — KPC000154 400mg Tablet administered orally in the morning once daily for 1 day
  Arms: KPC000154 400mg Tablet Intervention
Drug: KPC000154 80mg multiple-dose Tablet Intervention（To Be Determined） — KPC000154 80mg tablet administered orally in the morning for 14 days
  Arms: KPC000154 80mg multiple-dose Tablet Intervention（To Be Determined）
Drug: KPC000154 120mg multiple-dose Tablet Intervention（To Be Determined） — KPC000154 80mg tablet administered orally in the morning for 14 days
  Arms: KPC000154 120mg multiple-dose Tablet Intervention（To Be Determined）
Drug: KPC000154 40mg multiple-dose Tablet Intervention（To Be Determined） — KPC000154 120mg tablet administered orally in the morning for 14 days
  Arms: KPC000154 40mg multiple-dose Tablet Intervention（To Be Determined）
Drug: Placebo-controlled（SAD） — A placebo used in a single-dose study where participants receive either the experimental drug or the placebo.
  Arms: Placebo (SAD)
Drug: Placebo-controlled（MAD） — A placebo used in a multiple-dose study where participants receive either the experimental drug or the placebo.
  Arms: Placebo (MAD）

SUMMARY:
A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of KPC000154 Tablets in Healthy Subjects

DETAILED DESCRIPTION:
KPC000154 is a thyroid hormone receptor beta (THR-β) agonist that improves NASH by increasing hepatic fat metabolism and reducing fat toxicity. Preclinical studies have shown that KPC000154 significantly reduces lipid levels and liver fibrosis in animal models.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must fully understand the purpose, nature, procedures of the trial, and potential adverse reactions, and voluntarily participate as subjects, signing an informed consent form prior to the commencement of any study procedures.
2. Healthy male and female subjects aged 18 to 55 years (inclusive of boundary values), with multiple-dose administration trials requiring subjects to have low-density lipoprotein cholesterol (LDL-C) levels that are either close to or at the borderline elevation (i.e., 2.8 mmol/L (110 mg/dL) ≤ LDL-C < 4.1 mmol/L (160 mg/dL)) are eligible for inclusion.
3. Male subjects must weigh ≥ 50.0 kg, and female subjects ≥ 45.0 kg; single-dose administration trials require a body mass index (BMI) within the range of 19.0-26.0 kg/m² (inclusive of boundary values), while multiple-dose administration trials require a BMI within the range of 19.0-30.0 kg/m² (inclusive of boundary values).
4. Subjects must utilize effective contraceptive measures during the trial period and for six months after the last administration of the investigational drug, and must not plan to conceive, donate sperm, or donate ova.
5. Subjects must be capable of effective communication with the investigators and understand and comply with all requirements of this study.

Exclusion Criteria:

1. Individuals with an allergic constitution (e.g., known allergies to two or more medications or foods), or a history of allergies to KPC000154 or related excipients.
2. Individuals with acute illnesses occurring within two weeks prior to screening.
3. Individuals who have used any medication (including prescription drugs, over-the-counter drugs, traditional Chinese medicine preparations, and herbal remedies), health supplements, or functional vitamins within two weeks prior to screening.
4. Individuals who have used inhibitors or inducers of CYP3A4, CYP2B6, CYP2C8, CYP2C9, or BCRP within one month prior to screening (e.g., inducers-rifampicin, phenobarbital, carbamazepine, phenytoin; inhibitors-itraconazole, voriconazole, tenofovir, ketoconazole, azithromycin, amiodarone, verapamil, sertraline, perphenazine, thioridazine, dapsone, montelukast, quercetin, phenformin, sulfamethoxazole, tinidazole, clarithromycin, ritonavir, gemfibrozil, clopidogrel, fluconazole, icatibant, aspergillus fumigatus toxin C, neomycin, sulfasalazine, curcumin, elvitegravir, cyclosporine A).
5. Individuals with a history of chronic or severe diseases affecting the cardiovascular, liver, kidney, respiratory, hematopoietic, lymphatic, endocrine, immune, psychiatric, neurological, or gastrointestinal systems, or individuals with gastrointestinal, liver, kidney, or thyroid diseases that could affect drug absorption or metabolism within one year prior to screening.
6. Individuals with a history of photosensitivity, or those currently undergoing antibiotic treatment for acne, or those with a history of or currently suffering from immunodeficiency diseases, lupus erythematosus, or immune dysfunction.
7. Individuals with abnormal clinical significance in physical examination, vital signs, clinical laboratory tests (blood biochemistry tests with ALT > 1.5 times ULN, or AST > 1.5 times ULN, or total bilirubin > 1.5 times ULN), chest X-ray, cardiac ultrasound (only for multiple-dose trials), abdominal ultrasound (liver, gallbladder, spleen, pancreas, kidneys), and electrocardiogram, as assessed by the investigator (Note: In multiple-dose trials, blood biochemistry tests showing borderline elevations in total cholesterol and triglycerides do not constitute clinically significant abnormalities, i.e., total cholesterol < 6.2 mmol/L (240 mg/dL), triglycerides < 3.4 mmol/L (300 mg/dL)).
8. Individuals who cannot abstain from consuming beverages and foods containing caffeine or alcohol (including chocolate, tea, coffee, cola, etc.), or grapefruit, grapefruit products, dragon fruit, mango, pomelo, orange, starfruit, guava, etc., which affect drug metabolism, or individuals who cannot stop smoking from 48 hours before dosing until the end of the trial.
9. Individuals with prolonged QTc interval on ECG at screening: males with QTcF > 450 ms or females with QTcF > 470 ms (corrected by Fridericia's formula, calculated as QTcF = QT/(RR^0.33)).
10. Individuals with glomerular filtration rate (GFR) < 90 mL/min (calculated using the simplified MDRD formula: males: eGFR = 186 × creatinine (mg/dL)^(-1.154) × age^(-0.203); females: eGFR = 186 × creatinine (mg/dL)^(-1.154) × age^(-0.203) × 0.742); Note: creatinine units are mg/dL, and creatinine results in μmol/L must be converted to mg/dL for calculation, 1 μmol/L = 0.01131 mg/dL.
11. Individuals with any disease that increases the risk of gastrointestinal bleeding, such as acute gastritis or gastric and duodenal ulcers.
12. Individuals who have undergone major surgical procedures within six months prior to screening (excluding diagnostic surgeries), or those planning to undergo surgery during the study, or those who have undergone surgeries judged by the investigator to affect drug absorption, distribution, metabolism, or excretion.
13. Individuals who have received any vaccinations within four weeks prior to screening, or those planning to receive any vaccinations during the trial.
14. Individuals who have participated in other clinical trials within three months prior to screening (Note: the end time is defined as the last date of participation in the clinical trial).
15. Individuals who have engaged in blood donation within three months prior to screening, or those who have experienced blood loss (excluding menstrual blood loss) totaling 400 mL or more within six months prior to screening.
16. Individuals with a history of alcohol consumption, i.e., an average weekly intake exceeding 2 units of alcohol (1 unit = 360 mL of beer or 45 mL of liquor with 40% alcohol content or 150 mL of wine) within one year prior to screening, or those who cannot abstain from alcohol during the trial, or those with alcohol breath test results > 0.0 mg/100 mL.
17. Individuals with an average daily smoking rate exceeding 5 cigarettes within three months prior to screening, or those with positive cotinine urine tests.
18. Individuals with a history of drug abuse (including non-medical use of various anesthetics and/or psychotropic drugs) within one year prior to screening, or those with positive drug abuse screening (including morphine, methamphetamine, ketamine, ecstasy (MDMA), marijuana (THC), etc.).
19. Individuals who cannot tolerate venipuncture/indwelling catheters, or those with difficulties in blood collection, or those with a history of fainting at the sight of blood.
20. Individuals with swallowing difficulties, or special dietary requirements, who cannot accept uniform diets.
21. Individuals with hereditary fructose intolerance or glucose/galactose absorption disorders, or those with sucrose-isomaltase deficiency.
22. Individuals deemed by the investigator to have other conditions unsuitable for inclusion.
23. Female subjects who have used oral contraceptives within 30 days prior to screening.
24. Female subjects who have used long-acting estrogens or progestins (including progesterone-releasing intrauterine devices) or implant contraceptives within six months prior to screening.
25. Female subjects who have engaged in unprotected sexual intercourse with partners within 14 days prior to screening.
26. Female subjects with positive pregnancy tests or test results outside the normal range or not within the non-pregnant state range.
27. Pregnant or lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-03-07 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic profile of KPC000154 after single and multiple oral administration (Cmax) | 12.8 month
  Maximum plasma concentration (Cmax) of KPC000154
Pharmacokinetic profile of KPC000154 after single and multiple oral administration (AUC0-t) | 12.8 month
  Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC0-t) of KPC000154
Pharmacokinetic profile of KPC000154 after single and multiple oral administration (Tmax) | 12.8 month
  Time to reach maximum plasma concentration (Tmax) of KPC000154

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 12.8 month
  safety measures

CONTACTS AND LOCATIONS:
Locations (1):
- No.49, Huayuan North Road, Haidian District, Beijing City, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: December 25, 2024 (start date)--January 12, 2026(end date)

REFERENCES:
- [Result] https://cmab.yiigle.com/uploads/guide_html/%E9%9D%9E%E9%85%92%E7%B2%BE%E6%80%A7%E8%84%82%E8%82%AA%E6%80%A7%E8%82%9D%E7%97%85%E9%98%B2%E6%B2%BB%E6%8C%87%E5%8D%97(2018%E6%9B%B4%E6%96%B0%E7%89%88).html
- [Result] Osaki Y, Takasawa M, Doi K, Nishimura H, Iwaki T, Imaizumi M, Oku N, Hatazawa J, Kubo T. Auditory and tactile processing in a postmeningitic deaf-blind patient with a cochlear implant. Neurology. 2006 Sep 12;67(5):887-90. doi: 10.1212/01.wnl.0000234141.72891.13. PMID 16966560
- See also: Guidelines for the prevention and treatment of non-alcoholic fatty liver disease — https://cmab.yiigle.com/uploads/guide_html/%E9%9D%9E%E9%85%92%E7%B2%BE%E6%80%A7%E8%84%82%E8%82%AA%E6%80%A7%E8%82%9D%E7%97%85%E9%98%B2%E6%B2%BB%E6%8C%87%E5%8D%97(2018%E6%9B%B4%E6%96%B0%E7%89%88).html